CLINICAL TRIAL: NCT06728761
Title: Evaluation of the Impact of Calvados ("Trou Normand") Consumption on Gastric Emptying After a High-calorie Meal
Brief Title: Gastric Emptying With Trou Normand
Acronym: GASTON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 69HCL24_0480
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteer
Keywords: gastric emptying; calvados
MeSH Terms: interventions — Appetite

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calvados (Experimental): Ingestion of test drink: Calvados. The volunteer will be invited to drink 2.5 cl of Calvados 40° at the 70th minute of the meal, before the cheese and dessert
  Interventions: Behavioral: Standardised test meal; Behavioral: Ingestion of test drink; Diagnostic Test: Ultrasound measurement of the antral area; Diagnostic Test: Breathalyser for measurement of the level of exhaled ethanol; Behavioral: Discomfort; Behavioral: Appetite; Diagnostic Test: Pregnancy urine test carried out during the intake visit on the day of the protocol
- Water (Active Comparator): Ingestion of Control drink: Water. The volunteer will be invited to drink 2.5 cl of water at the 70th minute of the meal, before the cheese and dessert
  Interventions: Behavioral: Standardised test meal; Behavioral: Ingestion of Control drink; Diagnostic Test: Ultrasound measurement of the antral area; Diagnostic Test: Breathalyser for measurement of the level of exhaled ethanol; Behavioral: Discomfort; Behavioral: Appetite; Diagnostic Test: Pregnancy urine test carried out during the intake visit on the day of the protocol

INTERVENTIONS:
Behavioral: Standardised test meal — Ingestion of a 1850 Kcal standardised 'Christmas meal' identical for each session. It will consist of the following elements Assortment of Picard Mini-Puff Pastry Aperitifs: 70g = 210 Kcal 1 glass of white wine = 85 Kcal with the aperitif
  1 slice of vacuum-packed foie gras = 50 g = 230 Kcal
  1 portion of turkey leg 200 g = 250 Kcal 50 g turkey cream = 130 Kcal
  1 portion of steamed potatoes = 200 g = 160 Kcal
  1 glass of red wine = 85 Kcal to accompany the main course
  1 slice of white bread (30 g) = 55 Kcal to eat with the main course Blind test or control drink (trou normand or placebo = water) / 1 scoop of apple sorbet
  1 portion 30 g camembert = 90 Kcal + White bread 1 slice (30 g) = 85 Kcal with the cheese
  1 portion crumble 100 g = 250 Kcal The different elements will be weighed for each participant.
Behavioral: Ingestion of test drink — Ingestion of 2,5 cl Calvados 40° at the 70th min of the meal (before cheese and dessert)
  Arms: Calvados
Behavioral: Ingestion of Control drink — Ingestion of 2,5 cl water at the 70th min of the meal (before cheese and dessert)
  Arms: Water
Diagnostic Test: Ultrasound measurement of the antral area — Ultrasound measurement of the antral area in the volunteers lying in the 45° semi-recumbent position using an ultrasound machine (Venue Go™, GE Healthcare, Chicago, IL, USA) fitted with an abdominal transducer (probe C1-5, 1.5 to 5 MHz) to obtain a sagittal cross-section of the antrum in a plane including the left lobe of the liver and the aorta. This will be performed during the intake visit, immediately before the test drink ingestion (70th min of the meal) and 15, 45, 60, 90, 120, 150, 180 min after the end of the meal
Diagnostic Test: Breathalyser for measurement of the level of exhaled ethanol — Breathalyser performed during the intake visit, and 15, 90, 180 and 300 min (if the exhaled alcohol level measured at 180 minutes was greater than 0.25 mg/l of breath) after the end of the meal.
Behavioral: Discomfort — discomfort will be assessed using seven-choice Likert scales immediately before the test drink ingestion and 90 min and 180 min after the end of the standardized meal.
Behavioral: Appetite — Appetite will be assessed using seven-choice Likert scales immediately before the test drink ingestion and 90 min and 180 min after the end of the standardized meal.
Diagnostic Test: Pregnancy urine test carried out during the intake visit on the day of the protocol — Pregnancy urine test carried out during the intake visit on the day of the protocol for exclusion of pregnant woman.

SUMMARY:
In France, alcohol is responsible for 30% of road deaths. The risk of being responsible for a fatal accident is multiplied by 17.8 for drink-drivers, and accidents involving alcohol consumption are more serious than others: the number of people killed per 100 injured in hospital is 23 for accidents involving alcohol, compared with 10 for accidents without alcohol. Alcohol is therefore responsible for an increased risk of road accidents, resulting in a high rate of alcohol-impaired victims being treated in emergency departments and operating theatres. Their management is all the more difficult in the operating theatre because these victims have a high gastric content, increasing the risk of pulmonary inhalation of gastric contents during the general anaesthesia required to treat trauma. Inhalation is one of the main causes of anaesthesia-related mortality.

ccident rates are higher during the festive season. Drinking high-alcohol beverages is reputed to help the digestion of rich meals and therefore improve digestive tolerance (abdominal symptoms: heaviness, bloating) and appetite during festive meals. The 'trou normand' consists of drinking calvados (alcohol: 40°) + 1 scoop of sorbet during the meal to improve digestion. The 'trou normand' is very popular on social networks and on restaurant menus, particularly during festive occasions such as weddings and Christmas meals. This belief may encourage the consumption of strong alcohol during festive meals, which is added to the usual alcohol consumption during this type of meal (wine), significantly increasing blood alcohol levels since 2.5 cl of an alcoholic beverage at 40° will have the same effect as 10 cl of wine at 10-12°. However, the alleged benefit of alcohol consumption on gastric emptying has never been demonstrated. On the contrary, some data in the literature suggest that alcohol consumption is associated with a slowing of gastric emptying.

The aim of this study is therefore to evaluate specifically the effect of strong alcohol consumption on gastric emptying of the liquid and solid components of a festive meal, as well as the effect on abdominal symptoms and appetite.

After verification of eligibility criteria and gastric content by an initial ultrasound examination and an alcohol test, the volunteers will be asked to consume a standardised meal of 1850 Kcal accompanied by a 12 cl glass of white wine (12°) at the start of the meal, a 12 cl glass of red wine with the main course (12°) and 2 glasses of water (20 cl) over 90 minutes. According to the randomisation, the volunteer will be invited, before the cheese and dessert, at the 70th minute, to drink 2.5 cl of water + 1 scoop of sorbet or 2.5 cl of Calvados 40° + 1 scoop of sorbet before the cheese and dessert, which will then be consumed within 20 minutes.

Immediately before ingesting the test drink, an ultrasound examination of the antrum will be carried out to measure the antral cross-sectional area. An antral ultrasound will be carried out 15, 45, 60, 90, 120, 150 and 180 minutes after the end of the meal, blind to the drink ingested, and a breathalyser test will be carried out at times 15, 90, 180 min and possibly 300 min after the end of the meal if the exhaled alcohol level measured at 180 min was greater than 0.25 mg/l of exhaled air. Volunteers will also be asked to indicate their abdominal discomfort and appetite on a seven-choice Likert scale before starting to eat the meal, then at the end of the standardised meal, then 1 h 30 and 3 h after the end of the meal.

ELIGIBILITY:
Inclusion Criteria:

* adult volunteers ≥ 18 years and < 65 years of age
* with no significant medical history (American Society of Anesthesiologists class ASA 1)
* fasted for at least 6 hours for alcohol and solids
* signed informed consent
* affiliated to the social security system.

Exclusion Criteria:

* adults of full age under legal protection (guardianship, curatorship)
* young drivers holding a probationary licence
* persons deprived of their liberty by a judicial or administrative decision
* persons under psychiatric care
* a history of oeso-gastro-duodenal surgery
* current pregnancy or breast-feeding
* any pathology that may affect gastric volume: insulin-dependent diabetes or diabetes mellitus, gastro-oesophageal reflux, hypothyroidism or hyperthyroidism
* treatments affecting gastric motility (erythromycin, metoclopramide, etc.)
* any treatment incompatible with alcohol consumption
* any pathology incompatible with alcohol consumption (liver or neurological pathologies in particular)
* obesity defined by a body mass index ≥ 30 kg/m².
* Alcohol dependence (AUDIT questionnaire): Alcohol Use Disorders Identification Test) is a simple 10-question test.
* Volunteers with a direct hierarchical link to the investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
gastric emptying half-time of a standardised meal during the two sessions (calvados or water). | half-time of gastric emptying of the standardised will be calculated based on the measurement of the antral area performed 15, 45, 60, 90, 120, 150 and 180 minutes after the end of the standardised meal (1850 Kcal), blindly to the drink ingested
  determination of the half-time of gastric emptying of a standardised meal (1850 Kcal) based on repeated measurements of the antral surface after the end of the standardised meal in both sessions.

SECONDARY OUTCOMES:
gastric emptying rate during the two sessions | Calculation will be made based on ultrasound measurements of the antral area at 15 minutes and 90 minutes minutes after the end of the standardized meal
  gastric emptying rate based on ultrasound measurements of the antral area taken at 15 minutes and 90 minutes after the end of the standardized meal
discomfort and appetite | 90 min and 180 min after the end of the standardized meal
  discomfort and appetite will be assessed using seven-choice Likert scales immediately before the test drink ingestion and 90 min and 180 min after the end of the standardized meal Kikert scales 1 to 7. 7 is strong desire for food, high appetite
level of exhaled ethanol | Breathalyser during the intake visit, and 15, 90, 180 and 300 min (if the exhaled alcohol level measured at 180 minutes was greater than 0.25 mg/l of breath) after the end of the meal.
  Breathalyser for measurement of the level of exhaled ethanol

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Femme Mère enfant, Bron, Rhone, France

IPD SHARING:
Plan to Share IPD: No